CLINICAL TRIAL: NCT06539858
Title: Investigation of the Effect of Massage Application on Functional Status and Depression in Mothers in the Early Postpartum Period
Brief Title: Investigation of the Effect of Massage Application on Functional Status and Depression in Postpartum Mothers
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, ZEYNEP İCLAL SAG, research assisstant, University of Yalova
Other Study IDs: 2024/3
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Depression, Post-Partum; Massage; Functional Status
MeSH Terms: conditions — Depression, Postpartum | interventions — Massage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interventional group: This group will receive massage once a week for 4 weeks.
  Interventions: Other: massage
- non-intervention group: No intervention will be made to this group

INTERVENTIONS:
Other: massage — General back massage from the base of the neck to the sacrum. Classical massage techniques such as stroking and kneeding will be applied. To be performed by a specialist physiotherapist.
  Groups: Interventional group

SUMMARY:
Postpartum depression is a condition with high morbidity in mothers and negatively affects all family relationships. It has been observed that depression in the mother at only 2 months of age negatively affects the relationship between the baby and the mother, and that mothers who are depressed and therefore their babies feel more negatively. Symptoms usually start to appear from the 2nd or 3rd week after birth. At the same time, most people focus on the physical characteristics of the mother after birth, such as her reproductive system, while ignoring her full functionality. Full functionality is a multidimensional concept that includes personal care, baby care, family care, social and professional activities. In the first weeks after discharge, the functional status of the mother may differ as a result of the roles she assumes at home. Since the breastfeeding period will begin in new mothers, different treatment methods are preferred instead of drug treatment, one of which is massage therapy. It is thought that massage therapy relaxes the muscles and changes psychological factors. Previous studies conducted on postpartum women show that massage has a positive and healing effect on mothers. While previous studies frequently mention its effects on depression, it has also been observed that there are few studies mentioning its functional status. In light of this information, the aim of this study is to investigate the effects of massage on functional status and depression in postpartum women. For this purpose, there will be 2 groups randomized as intervention and control groups. The intervention will be performed as a 45-minute massage once a week for 4 weeks. Data will be collected before the first intervention and after the last intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being within the first 6 months postpartum

Exclusion Criteria:

* Having a health condition that prevents lying face down (having stitches from a cesarean section, hypertension, etc.)
* Not being cooperative
* All conditions that contraindicate massage

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young mothers who had just given birth and met the inclusion criteria for the study
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
depression | 4 weeks
  will be evaluated with the internationally accepted Edinburgh Postpartum Depression Scale. the name of the scale we use Edinburgh Postpartum Depression Scale. As the score obtained from this scale increases, the person's depression level also increases.
functionality | 4 weeks
  The change in functionality will be evaluated using the postpartum functional status inventory. Inventory of Functional Status After Childbirth Turkish was used. According to this scale, a decrease in the score indicates that the functional status also decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No